CLINICAL TRIAL: NCT04562441
Title: AXEL: Axitinib-Avelumab Combination in Recurrent or Metastatic Nasopharyngeal Cancer: a Multicenter Phase 2 Trial
Brief Title: NPC - AXEL Study : Axitinib-Avelumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Edwin P Hui, Director, CCTU, Department of Clinical Oncology, CUHK, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC 033
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Recurrent or Metastatic NPC
MeSH Terms: conditions — Recurrence | interventions — Axitinib; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axitinib and Avelumab (Experimental): Axitinib: 5 mg bd po Day 1 to Day 28
  Avelumab: 10mg/kg Day 1 and Day 15 every 4 weeks
  Interventions: Drug: Axitinib; Drug: Avelumab

INTERVENTIONS:
Drug: Axitinib — Axitinib: 5 mg bd po Day 1 to Day 28
Drug: Avelumab — Avelumab: 10 mg/kg Day 1 to Day 15 every 4 weeks

SUMMARY:
Nasopharyngeal cancer (NPC) is the most common head and neck cancer in South China and South East Asia. Worldwide, there are 80,000 incident cases and 50,000 deaths annually. In Hong Kong, NPC ranked as the tenth most common cancer in man. Up to 30% of NPC patients will develop recurrence or metastases after primary radiotherapy or chemoradiation. Platinum-based chemotherapy regimen has been the main stay of first line treatment for recurrent or metastatic NPC. However, the duration of response is short and currently there is no recommended standard second line chemotherapy. Axitinib is a highly potent and selective inhibitor of VEGF receptor. Selectively targeting a single growth factor receptor pathway provides the potential to rationally adjust dosages and combine drugs directed at specific parts of the pathway to minimize toxicity and achieve the optimum therapeutic benefit. In the phase 2 axitinib monotherapy in recurrent or metastatic NPC who failed at least one line of chemotherapy, the clinical benefit rate (CBR, complete response + partial response + stable disease) was 78.4% at 3 months but decreased to 43.2% at 6 months. However, the confirmed objective response rate (ORR) by RECIST was only 2.7% and unconfirmed ORR of 18.9%, with no complete response.Recently, the promising clinical activity of immune check point inhibitors has been demonstrated in NPC. The ORR was 25.9% (7 partial responses out of 27 patients) for single agent pembrolizumab, and 20.5% (including 1 complete response and 7 partial responses out of 44 patients) for single agent nivolumab,9 in recurrent or metastatic NPC who failed at least first line chemotherapy.

The combination of axitinib and avelumab has been studied in renal cell carcinoma (RCC). Based on the above promising and positive results in renal cell carcinoma (RCC) and head and neck squamous cell carcinomas (HNSCC), the investigators hypothesize that the combination of axitinib and avelumab in the second line setting of NPC will achieving a more complete, deep and durable response than either agent alone, without a significant increase in toxicity.

This is an open-label, single arm, phase 2 clinical trial evaluating the activity and safety of the combination of axitinib and avelumab in recurrent or metastatic NPC patients who failed at least one line of platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of nasopharyngeal carcinoma (NPC) (either at initial diagnosis or at recurrence).
* Available fresh or archival tumor tissue for biomarker study
* Patients with recurrent or metastatic NPC that has progressed following one line of prior platinum-based chemotherapy.
* Disease must be not amenable to potentially curative radiotherapy or surgery.
* At least one measurable lesion as defined by RECIST v1.1 that has not been previously irradiated.
* Age 18 or above;
* ECOG performance 0 or 1.
* Adequate bone marrow, renal and hepatic reserve.

Exclusion Criteria:

* Prior therapy with immune check point inhibitors or VEGF pathway inhibitors.
* Presence of local recurrence.
* Presence of neck lymph node recurrence invading vascular structure.
* Presence of central lung lesions involving major blood vessels.
* History of hemoptysis or epistaxis within 4 weeks.
* Preexisting uncontrolled hypertension defined as more than 140/90 mmHg despite adequate medical therapy.
* Gastrointestinal abnormalities, including inability to take oral medication or malabsorption syndrome.
* Concurrent use or anticipated need for treatment with known potent CYP3A4 inhibitors or CYP3A4 /CYP1A2 inducers.
* CNS metastases requiring systemic steroid
* Active autoimmune disease
* Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Confirmed objective response rate (ORR) | 2 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years
6-month PFS rate | 6 months
Overall survival (OS) | 3 years
OS rates at 12 months and 24 months | 2 years
Objective tumor response rate | 2 years
Disease control rate (DCR) at 12 and 24 weeks | 2 years
Time to tumor response (TTR) | 2 years
Duration of response (DR) | 2 years
Patient-Reported Outcomes (FACT-NP) | 2 years
Patient-Reported Outcomes (EQ-5D) | 2 years
Type, incidence, severity (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], Version 4.0) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Chan, MD, Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No